CLINICAL TRIAL: NCT05037084
Title: The Association Between Physical Behavior, Sleep and Neuropsychiatric Symptoms in Nursing Homes
Brief Title: Activity and Health in Nursing Homes
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Trondheim Kommune (Other)
Responsible Party: Sponsor
Other Study IDs: 157470
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Old Age; Frailty
Keywords: Nursing home; Physical activity
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
There is expected to be an increased need for full time nursing homes as the increase in number of older adults increases and the rate of dementia diagnosis happens simultaneous with the decrees of healthcare personnel the years to come. A lift in knowledge is needed to provide a better and more efficient healthcare to be better equipped to meet this societal challenge. Physical activity and sleep are important indicators of health, but also on effect of treatment and care for this frail population. Comprehensive mapping of personnel time spent on different tasks and older adults' physical function throughout a week gives a unique opportunity to gain new knowledge about everyday life in nursing homes. The main aim of this project is to describe associations between physical behavior, sleep and symptoms in residents in nursing homes in Trondheim Municipality and combine these with personnel time spent on different working tasks.

ELIGIBILITY:
Inclusion Criteria:

All residents in nursing homes in Trondheim Municipality.

Exclusion Criteria:

Terminal residents or residents that can not stand or walk a few steps independently.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All residents living full time in nursing homes. These are often frail older adults with reduced physical function, high number of medications and comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 1123 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Axivity accelerometer | 7 days
  Activity monitoring
Somnofy sleepmonitor | 7 days
  Sleep monitoring
Short Physical Performance Battery (SPPB) | Baseline
  Measurement of physical function

SECONDARY OUTCOMES:
Time register | 7 days
  Time used on different tasks during the work day
Neuropsychiatric Inventory (NPI) | Baseline
  provide a brief assessment of neuropsychiatric symptomatology in routine clinical practice settings
Dementia Staging Instrument (CDR) | Baseline
  characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Olsen, Study Chair — Trondheim Kommune
Locations (1):
- Trondheim Kommune, Trondheim, Norway